CLINICAL TRIAL: NCT01253889
Title: Glucose 25% and Facilitated Tucking for Reducing Procedural Stress During Neonatologist-performed Cardiac Echocardiography in Infants in the NICU
Brief Title: Sweetheart Study: Oral Glucose for Reducing Stress During Echocardiographic Assessment in Infants in the NICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Liisa Holsti, Tier 2 Canada Research Chair in Neonatal Health and Development, Children's & Women's Health Centre of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H10-02069
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Echocardiography Assessment
Keywords: Functional echocardiography; oral glucose; neonatal stress
MeSH Terms: interventions — Glucose; Solutions; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oral Glucose with soother (Active Comparator): Oral Glucose 25% first given two minutes before the first contact by the physician performing the np-ECHO. A soother will be held in the infant's mouth to ensure that continuous contact is maintained throughout the testing period. Repeat application of solution as per study protocol. No other non-pharmaceutical interventions for stress reduction will be applied. During each np-ECHO, infants have additional handling only if it is required to maintain physiological stability.
  Interventions: Drug: Glucose 25% oral solution
- Oral water with soother (Placebo Comparator): Oral water first given two minutes before the first contact by the physician performing the np-ECHO. A soother will be held in the infant's mouth to ensure that continuous contact is maintained throughout the testing period. Repeat application of solution as per study protocol. No other non-pharmaceutical interventions for stress reduction will be applied. During each np-ECHO, infants have additional handling only if it is required to maintain physiological stability.
  Interventions: Other: Oral water
- Oral glucose with soother and tucking (Active Comparator): For the infants randomized to receive facilitated tucking throughout the procedure, the bedside nurse will provide gentle, firm containment of the extremities. The facilitated tucking will commence immediately after the baseline BIIP score is taken, but before the glucose/water is administered.
  Interventions: Drug: Glucose 25% oral solution
- Oral water with soother and tucking (Placebo Comparator): For the infants randomized to receive facilitated tucking throughout the procedure, the bedside nurse will provide gentle, firm containment of the extremities. The facilitated tucking will commence immediately after the baseline BIIP score is taken, but before the glucose/water is administered.
  Interventions: Other: Oral water

INTERVENTIONS:
Drug: Glucose 25% oral solution — 0.5ml of 25% glucose (26-31 weeks gestational age group) or 1.0 ml of 25% glucose (32-42 weeks gestational age group). This application can be repeated if necessary to a maximum of four times, adding up to max 2ml of 25% glucose in the 26-31 weeks gestational age group or 4ml of 25% glucose in the 32-42 weeks gestational age group.
  Other Names: glucose
  Arms: Oral Glucose with soother; Oral glucose with soother and tucking
Other: Oral water — 0.5ml of oral water (26-31 weeks gestational age group) or 1.0 ml of oral water (32-42 weeks gestational age group). This application can be repeated if necessary to a maximum of four times, adding up to max 2ml of oral water in the 26-31 weeks gestational age group or 4ml of oral water in the 32-42 weeks gestational age group.
  Arms: Oral water with soother; Oral water with soother and tucking

SUMMARY:
The purpose of this study is to compare the effect of a 25% glucose solution given via a soother with or without facilitated tucking with a similarly administered water placebo (control condition) on infant stress responses during and immediately after a neonatologist performed ECHO (np-ECHO).

DETAILED DESCRIPTION:
One hundred and four infants were randomized to one of four groups during a single np-ECHO examination, at the discretion of the medical team. Randomization to soother and water (Control) with and without facilitated tucking or to soother and 25% glucose (Intervention) with or without facilitated tucking will be determined by generating randomly permuted sequential blocks of four and six allocation numbers.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 26-42 weeks of gestational age admitted to the Neonatal Intensive Care Unit who require a np-ECHO for clinical purposes as indicated by the medical team.

Exclusion Criteria:

* Infants who have congenital anomalies, or a lethal condition in whom intensive care is not indicated;
* Infants below the gestational age of 26 completed weeks;
* Infants who have received analgesics or sedatives within 72 hours of the assessment;
* History of maternal abuse of controlled drugs and substances.
* Infants who are too unstable to receive oral medications or be exposed to a np-ECHO or who already have had an ECHO performed by a Pediatric Cardiologist within 4 hours.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Indicators of Infant Pain (BIIP) Score | study day 1
  The Behavioral Indicators of Infant Pain (BIIP) is a reliable and valid scale for assessing acute procedural pain in preterm infants.

SECONDARY OUTCOMES:
Time to complete a standard ECHO | study day 1
  Defined when ultrasound images have been acquired for all four cardiac views
Total number of times solutions are given to infants (max 4 times) | study day 1
Quality of np-ECHO images assessed by blinded cardiologists | study day 1
Mean heart rate from baseline to end of ECHO | study day 1
Cardiorespiratory instability | study day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Children's & Women's Health Centre of BC, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Lavoie PM, Stritzke A, Ting J, Jabr M, Jain A, Kwan E, Chakkarapani E, Brooks P, Brant R, McNamara PJ, Holsti L. A Randomized Controlled Trial of the Use of Oral Glucose with or without Gentle Facilitated Tucking of Infants during Neonatal Echocardiography. PLoS One. 2015 Oct 23;10(10):e0141015. doi: 10.1371/journal.pone.0141015. eCollection 2015. PMID 26496361